CLINICAL TRIAL: NCT00717223
Title: A Survey To Elicit The Relationship Between Literacy And Glycemic Control In Pediatric Diabetes
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rubina Heptulla, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-21263
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 1 diabetes mellitus; Type 2 diabetes mellitus; Literacy; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Literacy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parents with children with diabetes: parents who have children 18 or younger with diabetes

SUMMARY:
The purpose of this study is to see if a patient's ability (and/ or parent) to read, write, and do basic math problems affects blood sugar control in children with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
"Literacy" is defined as an individual's ability to read, write, and speak English, and compute and solve problems at levels of proficiency necessary to function on the job and in society, to achieve one's goals, and develop one's knowledge and potential, according to the National Literacy Act of 1991. The National Work Group on Health and Literacy reported that between 40 and 44 million persons in the United States have rudimentary literacy skills, and are unable to understand written materials that require only basic reading proficiency. Illiteracy has become an increasingly important problem, especially as it relates to healthcare. Literacy skills are paramount to effective self-management of type 1 and type 2 diabetes mellitus. And, "Diabetes Self-Management Education" is the cornerstone of care for all individuals with diabetes who want to achieve successful health-related outcomes. Self care of diabetes plays a major role in achieving DCCT recommended level of hemoglobin A1C. Deficient self-management will lead to uncontrolled diabetes, resulting in multisystem complications, increasing exponentially the burden on our healthcare system. Structured education of individuals tailored to combat poor literacy skills is imperative in helping these individuals achieve good glycemic control. Hence we would like to evaluate literacy in our clinic so appropriate educational material can be developed to help patient with T1DM who have low literacy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus
* Parent/ legal guardian must be present if child is less than 18 years of age.
* Diagnosis of type 1 or type 2 diabetes mellitus must have been made at least 1 year earlier.
* Parent/ legal guardian and/ or child must have completed all 3 mandatory diabetes education classes.
* English and/or Spanish speaking only.

Exclusion Criteria:

* Any form of mental retardation or cognitive disorder in parent/ legal guardian.
* Mental retardation or cognitive disorder in a child who is in Grade 6 or higher.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with diabetes attending clinic followup at Texas Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Literacy levels and HbA1c | 1 year
  look at literacy levels an HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Diabetes Clinic, Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassan K, Heptulla RA. Glycemic control in pediatric type 1 diabetes: role of caregiver literacy. Pediatrics. 2010 May;125(5):e1104-8. doi: 10.1542/peds.2009-1486. Epub 2010 Apr 5. PMID 20368322